CLINICAL TRIAL: NCT05127057
Title: Proactive and Integrated Management and Empowerment in Parkinson's Disease (PRIME-UK): A New Model of Care
Brief Title: Proactive and Integrated Management and Empowerment in Parkinson's Disease (PRIME-UK): A New Model of Care (PRIME-RCT)
Acronym: PRIME-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bristol (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2020-7271
Record Dates: First submitted 2021-10-19; First posted 2021-11-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Parkinsonism
Keywords: Lewy body dementia; Idiopathic Parkinson's Disease; Multiple System Atrophy; Progressive Supranuclear Palsy; Corticobasal degeneration; Vascular dementia
MeSH Terms: conditions — Parkinsonian Disorders; Lewy Body Disease; Parkinson Disease; Multiple System Atrophy; Supranuclear Palsy, Progressive; Corticobasal Degeneration; Dementia, Vascular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRIME Parkinson Care (Experimental): PRIME Parkinson Care is a multi-component model of care comprising individual components: a) Case management b) Empowerment of patients and care givers c) Empowerment of healthcare professionals d) IT infrastructure.
  Interventions: Other: PRIME Parkinson Care; Other: Usual Care
- Usual care (Placebo Comparator): Usual care provided by NHS
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: PRIME Parkinson Care — A novel model of care
  Arms: PRIME Parkinson Care
Other: Usual Care — Usual NHS Care

SUMMARY:
People living with Parkinson's disease experience progressive motor and non-motor symptoms, which negatively impact on health-related quality of life. Symptoms emerge and evolve as the disease progresses.

Current care models are often inadequate to meet their needs.

This study aims to evaluate whether a complex and innovative model of integrated care will increase an individual's ability to achieve their personal goals, have a positive impact on health and symptom burden, and be more cost-effective when compared with usual care.

DETAILED DESCRIPTION:
Background: People living with Parkinson's disease experience progressive motor and non-motor symptoms, which negatively impact on health-related quality of life and can lead to an increased risk of hospitalisation. It is increasingly recognised that the current care models are not suitable for the needs of people with parkinsonism whose care needs evolve and change as the disease progresses. This study aims to evaluate whether a complex and innovative model of integrated care will increase an individual's ability to achieve their personal goals, have a positive impact on health and symptom burden, and be more cost-effective when compared with usual care.

Methods: This is a single centre, randomised controlled trial where people with parkinsonism and their informal caregivers are randomised into one of two groups: either PRIME Parkinson multi-component model of care; or usual care. Adults ≥18 years with a diagnosis of parkinsonism, able to provide informed consent or the availability of a close friend or relative to act as a personal consultee if capacity to do so is absent, and living in the trial geographical area are eligible. Up to three caregivers per patient can also take part, must be ≥18 years, provide informal, unpaid care and able to give informed consent. The primary outcome measure is goal attainment, as measured using the Bangor Goal Setting Interview. The duration of enrolment is 24 months. The total recruitment target is n=214 and the main analyses will be intention to treat.

Discussion: This trial tests whether a novel model of care improves health and disease-related metrics including goal attainment, and decreases hospitalisations whilst being more cost-effective than the current usual care. Subject to successful implementation of this intervention within one centre, the PRIME Parkinson model of care could then be evaluated within a cluster-randomised trial at multiple centres.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of parkinsonism made by a movement disorder specialist
2. Be willing to participate
3. Have the ability to provide informed consent to participant, or where unable to do so due to cognitive impairment, availability of a close friend or relative to act as a personal consultee
4. Age 18 years and above.
5. Resident within the geographical catchment area of Royal United Hospital Bath NHS Foundation Trust, UK

Exclusion Criteria:

1. Patients with drug, infection or toxin induced parkinsonism
2. Patients who lack capacity to participate but do not have anyone who can be a consultee to provide advice regarding the patient's wishes and views
3. Patients with a current medical, cognitive or psychosocial issue or co-enrolment in other study that, in the opinion of the site investigator, would interfere with adherence to study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Goal attainment | 24 months
  Measured using the Bangor Goal-Setting Interview (BGSI) - score 1-10, higher score = better outcome

SECONDARY OUTCOMES:
Parkinson's disease assessment | 24 months
  Measured using MDS-Unified Parkinson's disease Rating Scale (MDS-UPDRS) Score range 0-199, higher score = worse outcome
Non-motor symptom burden | 24 months
  Measured using MDS-Non-motor rating scale (MDS-NMS); Score range 0-334, higher score = worse outcome
Parkinson's-related quality of life | 24 months
  Measured using The Parkinson's Disease Questionnaire (PDQ-39); Score range 0-100, higher score = worse outcome
Fear of falling | 24 months
  Measured using the Iconographical Falls Efficacy Scale (ICON-FES); Score range 10-40, higher score = worse outcome
Global Impression of change | 24 months
  Measured using the Patients' Global Impression of Change (PGIC);Score range 0-7, higher score = worse outcome
Frailty | 24 months
  Measured using The Frailty Instrument of the Survey of Health, Ageing and Retirement in Europe (SHARE-FI75+); Score range 0-1, higher score = worse outcome. Measured using Measured using Pictorial fit frail scale; Score range 0-43, higher score = worse outcome. Measured using clinical frailty scale; Score range 0-9, higher score = worse outcome
Sarcopenia | 24 months
  Measured using the Sluggishness, Assistance in walking, rising from a chair, climb stairs, falls questionnaire (SARC-F); Score range 0-10, higher score = worse outcome
Malnutrition risk | 24 months
  Measured using the Malnutrition Universal Screening Tool (MUST); Score range 0-6, higher score = worse outcome. Measured using the Seniors in the community: risk evaluation for eating and nutrition (SCREEN-II-14); Score range 0-64, higher score = better outcome.
Physical performance | 24 months
  Measured using the Short Physical Performance Battery (SPPB); Score range 0-12, higher score = better outcome. Measured using the Timed up and Go (TUG); score is not a scale (timing).
Physical activity | 24 months
  Measured using the Incidental and Planned Exercise Questionnaire - WA Version (IPEQ-WA); Score range 0-182, higher score = better outcome
Gait | 24 months
  Measured using single and dual task gait assessments
Grip strength | 24 months
  Measured using hand-held dynamometer; scoring is in kg not a scale
Advance Care Plan data | 24 months
  Measured using the Edmonton Symptom Assessment System - Revised: Parkinson's disease (ESAS-R-PD); Score range 0-100, higher score = worse outcome
Palliative symptom burden | 24 months
  Measured using the Palliative Case Outcome Scale - symptom list: Parkinson's disease (POS-S-PD); Score range 0-40, higher score = worse outcome
Hospice utilisation outside place of death | 24 months
  Captured from hospital and GP records
Use of anticipatory medication | 24 months
  Captured from hospital and GP records
Healthcare contacts with hospice and/or palliative care services | 24 months
  Captured from hospital and GP records
Loneliness/social isolation | 24 months
  Measured using UCLA-Loneliness Scale (3-item); Score range 3-9, higher score = worse outcome
Social participation | 24 months
  Measured using the English Longitudinal Study of Ageing questionnaire (ELSA) - scoring not a scale
Perceived social support | 24 months
  Measured using Multidimensional scale of perceived social support (MSPSS); Score range 12-84, higher score = better outcome
Coping strategy | 24 months
  Measured using the Brief Coping Orientation to Problems Experienced Inventory (BRIEFCope); Score range 28-112, higher score = better outcome
Acceptance of illness | 24 months
  Measured using Acceptance of Illness Scale; Score range 8-40, higher score = better outcome
Capability | 24 months
  Measured using the ICEpop Capability measure for older people (ICECAP-O); Score range 5-20, higher score = better outcome
Patient Activation | 24 months
  Measured using Patient Activation Measure (PAM); Score range 0-100, higher score = better outcome
Health related quality of life | 24 months
  Measured using EuroQol 5D-5L (EQ-5D-5L); Score range 5-25, higher score = worse outcome
Mortality | 24 months
  Captured from hospital and GP records
Healthcare events | 24 months
  Captured from hospital and GP records
Frequency of Parkinson's follow-up | 24 months
  Captured from hospital and GP records
Frequency and type of engagement with PRIME Parkinson care | 24 months
  Captured from study information
Experience of holistic patient-centred care | 24 months
  Measured using Patient Assessment of Chronic Illness Care (PACIC-26); Score range 26-130, higher score = better outcome
Montreal Cognitive Assessment | 24 months
  Measured using Montreal Cognitive Assessment
Bone health | 24 months
  Measured using a combination of QFracture and FRAX questionnaires
Life space assessment | 24 months
  Measured using LSA questionnaire collecting participant's movements over the last month

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Henderson, PhD, Principal Investigator — University of Bristol
Locations (1):
- Population Health Sciences, University of Bristol, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lloyd K, Tenison E, Smith S, Lithander F, Kidger J, Brant H, Redwood S, Ben-Shlomo Y, Henderson EJ. Exploring how PRIME-Parkinson care is implemented and whether, how and why it produces change, for who and under what conditions: a protocol for an embedded process evaluation within the PRIME-UK randomised controlled trial. BMJ Open. 2025 Feb 2;15(1):e086353. doi: 10.1136/bmjopen-2024-086353. PMID 39894518